CLINICAL TRIAL: NCT04638751
Title: ARGONAUT: Development and Analysis of a Blood and Stool Sample Bank for Cancer Patients, Enabling the Systematic Study of the Effect of Gut Microbiomes on Response to Treatment
Brief Title: ARGONAUT: Stool and Blood Sample Bank for Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Persephone Biosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: PB-2020-01
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Non-small Cell Lung Cancer; Colorectal Cancer; Triple Negative Breast Cancer; Pancreas Cancer
Keywords: microbiome; immunotherapy; checkpoint inhibitor; cancer; colonoscopy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Triple Negative Breast Neoplasms; Pancreatic Neoplasms; Neoplasms | interventions — Immunotherapy; Drug Therapy; Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- NSCLC: Stage 3 or stage 4 non-small cell lung cancer patients, being administered checkpoint inhibitor therapy for the first time. Dosage form, dosage, frequency and duration will be either standard of care and accessed via normal commissioning arrangements, or will be part of an ethics-approved clinical trial, where co-enrollment into an observational study is permitted.
  Interventions: Drug: Immunotherapy
- Triple-negative breast cancer: Stage 3 or stage 4 metastatic triple-negative breast cancer patients, being administered any type of treatment that the patient has not experienced before. Dosage form, dosage, frequency and duration will be either standard of care and accessed via normal commissioning arrangements, or will be part of an ethics-approved clinical trial, where co-enrollment into an observational study is permitted.
  Interventions: Drug: Chemotherapy
- Colorectal cancer: Stage 3 or stage 4 colorectal cancer patients, being administered any type of treatment that the patient has not experienced before. Dosage form, dosage, frequency and duration will be either standard of care and accessed via normal commissioning arrangements, or will be part of an ethics-approved clinical trial, where co-enrollment into an observational study is permitted.
  Interventions: Drug: Immunotherapy; Drug: Chemotherapy; Procedure: CRC surgical resection
- Pancreatic cancer: Stage 3 or stage 4 pancreatic cancer patients, being administered any type of treatment that the patient has not experienced before. Dosage form, dosage, frequency and duration will be either standard of care and accessed via normal commissioning arrangements, or will be part of an ethics-approved clinical trial, where co-enrollment into an observational study is permitted.
  Interventions: Drug: Immunotherapy; Drug: Chemotherapy
- High risk for colorectal cancer: Subjects undergoing a standard-of-care colonoscopy for colorectal cancer (CRC) screening considered at high risk for CRC due to either 1) one or more first degree relatives with a history of CRC, or 2) a personal history of colorectal cancer, advanced adenoma as defined by USMSTF guidelines on colorectal cancer, or 3 or more non-advanced adenomas in a single screening or surveillance encounter (synchronous).
  Interventions: Procedure: Colonoscopy
- Low risk for colorectal cancer: Subjects undergoing a standard-of-care colonoscopy for colorectal cancer (CRC) screening, who are not considered high risk for CRC based on family history or prior colonoscopy findings.
  Interventions: Procedure: Colonoscopy

INTERVENTIONS:
Drug: Immunotherapy — Checkpoint inhibitor
  Groups: Colorectal cancer; NSCLC; Pancreatic cancer
Drug: Chemotherapy — Any form of chemotherapy
  Groups: Colorectal cancer; Pancreatic cancer; Triple-negative breast cancer
Procedure: CRC surgical resection — Surgical resection to remove colorectal cancer
  Groups: Colorectal cancer
Procedure: Colonoscopy — Standard-of-care colonoscopy for CRC screening
  Groups: High risk for colorectal cancer; Low risk for colorectal cancer

SUMMARY:
ARGONAUT is a longitudinal, prospective, observational study that will enroll up to 5,000 advanced-stage cancer patients of diverse racial backgrounds to collect data used to develop precision microbiome medicines and for the identification of clinically actionable cancer-specific biomarkers to guide therapeutic decisions. Four types of solid tumor cancers will be profiled including non-small cell lung cancer (NSCLC), triple negative breast cancer (TNBC), colorectal cancer (CRC) and pancreatic cancer. Healthy control subjects without a cancer diagnosis will also be studied, comprised of individuals at high risk for CRC and healthy individuals at low risk for CRC. Risk assessment will be based on family history or past neoplastic findings during CRC screening. Data collected from this study will be used to develop the most effective new therapies, via microbiome optimization, all to the benefit of patients and the physicians treating them. Stool and blood samples will be collected longitudinally and analyzed to determine the impact of gut microbiome composition and function on the immune system and efficacy of the treatment.

Currently enrolling the CRC, high risk, and low risk cohorts.

Subjects who meet the entry criteria will provide up to 5 samples each of blood and stool over a 2-year period. Approximately 10%-20% of the subjects will provide colon tissue samples, either from research biopsies during Standard of Care (SOC) screening colonoscopy or retained surgical tissue from colectomy. Electronic health records will be obtained at various times for up to 8 years, to collect tumor imaging results and any other updated medical data, with no additional samples collected. In select cases, stool and blood samples will be collected beyond 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Men or women who are ≥ 18 years old with stage III or stage IV non-small cell lung cancer (NSCLC), colorectal cancer, triple-negative breast cancer, or pancreatic cancer treated by a particular cancer treatment for the first time, OR healthy subjects undergoing a standard of care colonoscopy
* Subjects able to provide written informed consent

Exclusion Criteria:

* Subjects with known HIV, Hepatitis A, Hepatitis B, Hepatitis C, or SARS-CoV2
* Subjects without the mental capacity to complete either a written or online questionnaire, alone or with assistance, or make sound decisions
* Women who are pregnant or who plan on becoming pregnant
* Women who are nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: It is anticipated that up to 5000 subjects will be enrolled in this study. It is preferred that enrollment is balanced by sex; however, it is not required. All efforts will be made to provide racial/ethnic balance, with a goal of 20% African American and 10% each of patients with Asian or Hispanic descent.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine whether the microbiome composition can predict progression-free survival | 6-12 months
  Whole genome sequencing and metabolomics will be used to characterize the patient's microbiome, and whether there is any correlation with response to treatment
Determine whether the microbiome composition can predict risk for colorectal cancer | 2-8 years
  Whole genome sequencing and metabolomics will be used to characterize the patient's microbiome. High and low risk subjects will be followed for 8 years to determine if any get CRC.

SECONDARY OUTCOMES:
Identify correlations between microbiome composition and immune markers | 6-12 months
  CyTOF and cytokine analysis will be performed on the blood samples to characterize the patient's immune phenotype
Determine whether the microbiome composition can predict overall survival | 6-24 months
  Survival and tumor progression will be monitored for an extended time beyond sample collection
Build a library of samples and data for future research | 6-24 months
  Samples will be stored and data saved in a HIPAA-compliant database. Samples will be linked to patient metadata.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Knowledge Research Center, Orange, California
  - SDG Clinical Research, Inc, San Diego, California
  - Persephone Biosciences, Inc., San Diego, California
  - L&A Morales Healthcare, Inc, Miami, Florida
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Mid-Hudson Medical Research, New Windsor, New York
  - Kroger Health, The Little Clinic, Cincinnati, Ohio
  - Southwest Family Medicine Associates, Dallas, Texas
  - Biopharma Informatic, Houston, Texas